CLINICAL TRIAL: NCT01937299
Title: Additive Effect of Brinzolamide 1%/Brimonidine 0.2% Fixed Dose Combination As Adjunctive Therapy to Travoprost
Brief Title: Effect of SIMBRINZA® Suspension as an Added Therapy to TRAVATAN Z®
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M-13-019
Record Dates: First submitted 2013-09-04; First posted 2013-09-09 (Estimated); Results first posted 2015-05-14 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-04

CONDITIONS: Ocular Hypertension; Open Angle Glaucoma
Keywords: glaucoma; prostaglandin analogue; brinzolamide; brimonidine
MeSH Terms: conditions — Ocular Hypertension; Glaucoma, Open-Angle; Glaucoma | interventions — brinzolamide; Brimonidine Tartrate; Travoprost; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SIMBRINZA (Experimental): Brinzolamide 1%/brimonidine 0.2% ophthalmic suspension, 1 drop in each eye 3 times a day (8 AM, 3 PM, 10 PM), with travoprost 0.004% ophthalmic solution, 1 drop in each eye at bedtime, for 6 weeks
  Interventions: Drug: Brinzolamide 1%/brimonidine 0.2% ophthalmic suspension; Drug: Travoprost 0.004% ophthalmic solution
- Vehicle (Placebo Comparator): Inactive ingredients, 1 drop in each eye 3 times a day (8 AM, 3 PM, 10 PM), with travoprost 0.004% ophthalmic solution, 1 drop in each eye at bedtime, for 6 weeks
  Interventions: Drug: Vehicle; Drug: Travoprost 0.004% ophthalmic solution

INTERVENTIONS:
Drug: Brinzolamide 1%/brimonidine 0.2% ophthalmic suspension
  Other Names: SIMBRINZA®
  Arms: SIMBRINZA
Drug: Vehicle — Inactive ingredients used as a placebo comparator
  Arms: Vehicle
Drug: Travoprost 0.004% ophthalmic solution
  Other Names: TRAVATAN Z®

SUMMARY:
The purpose of this study is to demonstrate the additive effect of brinzolamide 1%/brimonidine 0.2% (SIMBRINZA® suspension) in subjects with either open angle glaucoma or ocular hypertension who are currently on a prostaglandin analogue (PGA) monotherapy (TRAVATAN Z®).

DETAILED DESCRIPTION:
This study was divided into 2 sequential phases. The Screening/Eligibility Phase included one Screening Visit and two Eligibility Visits, during which subjects washed out of all other intraocular pressure (IOP)-lowering medications and dosed with TRAVATAN Z®, 1 drop instilled in each eye once daily for 28 days. Subjects who met all inclusion/exclusion criteria were randomized at the second Eligibility Visit. The Treatment Phase consisted of two on-therapy visits (Week 2 and Week 6).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of open angle glaucoma or ocular hypertension;
* Mean IOP measurements in at least 1 eye (study eye) of ≥ 21 mmHg and <32 mmHg at 8 AM while on travoprost monotherapy at 2 consecutive visits (Eligibility 1 and Eligibility 2);
* Able to understand and sign Informed Consent form;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Women of childbearing potential who are pregnant, breastfeeding, or do not agree to use an adequate birth control method throughout the study;
* Any form of glaucoma other than open angle glaucoma or ocular hypertension;
* Severe central visual field loss;
* Chronic, recurrent, or severe inflammatory eye disease;
* Ocular trauma within the past 6 months;
* Ocular infection or ocular inflammation within the past 3 months;
* Best-corrected visual acuity score worse than approximately 20/80 Snellen;
* Eye surgery within the past 6 months;
* Any condition, including severe illness, which would make the subject unsuitable for the study in the opinion of the Investigator;
* Use of any additional topical or systemic ocular hypertensive medication during the study;
* Patients who, in the opinion of the Investigator, cannot discontinue all IOP-lowering ocular medication(s) per the appropriate washout schedule prior to Eligibility 1 Visit;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2013-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Burmaster, PhD, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 32 investigational centers located in the US.
Pre-assignment Details: Of the 307 enrolled, 74 participants were exited as screen failures prior to randomization. This reporting group includes all randomized participants (233).
Groups:
- SIMBRINZA; Vehicle: 1 drop in each eye 3 times a day (8 AM, 3 PM, 10 PM), with travoprost 0.004% ophthalmic solution, 1 drop in each eye at bedtime, for 6 weeks
Period: Overall Study
Arm/Group | SIMBRINZA | Vehicle
Started | 117 | 116
Completed | 103 | 112
Not Completed | 14 | 4
Not completed — Adverse Event | 13 | 0
Not completed — Lack of Efficacy | 0 | 4
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all subjects who received study medication and completed at least 1 scheduled on-therapy study visit (intent-to-treat).
Groups:
- SIMBRINZA: 1 drop instilled 3 times a day in each eye for 6 weeks as adjunctive therapy to travoprost ophthalmic solution 0.004%
- Vehicle: 1 drop instilled 3 times a day in each eye for 6 weeks in conjunction with travoprost ophthalmic solution 0.004%
- Total: Total of all reporting groups
Arm/Group | SIMBRINZA | Vehicle | Total
Number analyzed (Participants) | 113 | 116 | 229
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (10.3) | 66.0 (10.6) | 66.8 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 67 | 136
  Male | 44 | 49 | 93
Mean Diurnal Intraocular Pressure (IOP) at Baseline [Mean (Standard Deviation); unit: mmHg] — Diurnal IOP at Baseline was defined as the average of the four Baseline IOP measurements at timepoints 8 AM, 10 AM, 3 PM, and 5 PM. For each timepoint, the baseline IOP was defined as the average of the timepoint-matched IOP measurements at the Eligibility 1 and Eligibility 2 Visits.
  mmHg | 22.48 (2.507) | 22.66 (2.407) | 22.57 (2.453)

OUTCOME MEASURES:

1. Primary Outcome: Mean Diurnal Intraocular Pressure (IOP) at Week 6
Description: Diurnal IOP was defined as the average of the four timepoints measured (8 AM, 10 AM, 3 PM, and 5 PM). IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry and reported in millimeters mercury (mmHg). One eye was chosen as the study eye and only data for the study eye were used for the analyses. A higher IOP can be a greater risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage).
Time Frame: Week 6
Population: This analysis population includes all subjects who received study medication and completed at least 1 scheduled on-therapy study visit. Last observation carried forward (LOCF) was not utilized; therefore results report subjects present at Week 6 with no imputation for missingness.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SIMBRINZA | Vehicle
Number analyzed (Participants) | 103 | 112
mmHg | 17.44 (2.838) | 20.34 (3.702)

2. Secondary Outcome: Mean Diurnal IOP Change From Baseline to Week 6
Description: Baseline IOP was defined as the average of the timepoint-matched IOP measurements at Eligibility 1 and Eligibility 2 Visits. Diurnal IOP change was defined as the average of the four changes from baseline (timepoints 8 AM, 10 AM, 3 PM, and 5 PM). IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry and reported in millimeters mercury (mmHg). One eye was chosen as the study eye and only data for the study eye were used for the analyses. A more negative change from baseline indicates a greater improvement, i.e., a reduction of IOP.
Time Frame: Baseline, Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SIMBRINZA | Vehicle
Number analyzed (Participants) | 103 | 112
mmHg | -5.10 (2.637) | -2.22 (2.925)

3. Secondary Outcome: Mean Diurnal IOP Percentage Change From Baseline to Week 6
Description: Baseline IOP was defined as the average of the timepoint-matched IOP measurements at Eligibility 1 and Eligibility 2 Visits. Diurnal IOP Percentage Change was defined as the average of the four percent changes from baseline (timepoints 8 AM, 10 AM, 3 PM, and 5 PM). IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry and reported in millimeters mercury (mmHg). One eye was chosen as the study eye and only data for the study eye were used for the analyses. A more negative percent change from baseline indicates a greater amount of improvement, i.e., a reduction of IOP.
Time Frame: Baseline, Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | SIMBRINZA | Vehicle
Number analyzed (Participants) | 103 | 112
percent change | -22.27 (10.842) | -9.57 (12.923)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study, Oct 2013-Apr 2014. This analysis population includes all consented subjects. Adverse events are reported as pre-treatment and treatment-emergent.
Description: An AE was defined as any untoward medical occurrence in a subject who was administered a study medication, regardless of whether or not the event had a causal relationship with the medication. All AEs were obtained as solicited and spontaneous comments from the subjects, and as observations by the Investigator, as outlined in the study protocol.
Groups:
- Pre-Treatment: Travoprost 0.004% ophthalmic solution, 1 drop in each eye at bedtime for a 4-week run-in period
- SIMBRINZA; Vehicle: 1 drop in each eye 3 times a day (8 AM, 3 PM, 10 PM), with travoprost 0.004% ophthalmic solution, 1 drop in each eye at bedtime for a 6-week treatment period
Arm/Group | Pre-Treatment | SIMBRINZA | Vehicle
Serious Adverse Events (participants affected / at risk) | 1/307 | 0/117 | 0/116
Other Adverse Events (participants affected / at risk) | 3/307 | 26/117 | 12/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-Treatment (N=307) | SIMBRINZA (N=117) | Vehicle (N=116)
Syncope (Nervous system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-Treatment (N=307) | SIMBRINZA (N=117) | Vehicle (N=116)
Conjunctival hyperaemia (Eye disorders) | 2 | 16 | 7
Vision blurred (Eye disorders) | 0 | 7 | 5
Dry mouth (Gastrointestinal disorders) | 1 | 9 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.